CLINICAL TRIAL: NCT03897543
Title: A Phase 1-2 Study of ABX196 in Combination With Nivolumab in Patients With Hepatocellular Carcinoma
Brief Title: ABX196 in Combination With Nivolumab in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Collaborators: C3 Research Associates (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX196-001
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; Nivolumab; ABX196
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ABX196

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABX196 (Experimental): IM injection of 0.1, 0.2, and 0.4 µg of ABX196
  Interventions: Drug: ABX196

INTERVENTIONS:
Drug: ABX196 — ABX196 will be administered as an IM injection 120 minutes (+/- 15 minutes) after the completion of the nivolumab infusion on Day 1 of every other 28-Day treatment cycle (i.e., every 8 weeks).

SUMMARY:
Open-label, uncontrolled, phase 1-2 study to evaluate the safety, tolerability, pharmacodynamic effects, and preliminary efficacy of ABX196 administered in combination with nivolumab in patients with hepatocellular carcinoma

DETAILED DESCRIPTION:
This is an open-label, uncontrolled phase 1-2 study to evaluate the safety, tolerability, pharmacodynamic effects, and preliminary efficacy of ABX196 administered in combination with nivolumab in patients with hepatocellular carcinoma. The study consists of 2 phases, a Dose Escalation Phase and an Expansion Phase. Nivolumab will be administered, consistent with the US prescribing information, as a 30-minute IV infusion on Days 1 and 15 of each 28-Day cycle. ABX196 will be administered as an IM injection 120 minutes (+/- 15 minutes) after the completion of the nivolumab infusion on Day 1 of every other 28-Day cycle (i.e., every 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Men or women, Age ≥18 years
* Patients with ECOG performance status 0 or 1
* Patients with histologically confirmed diagnosis of HCC not amenable to curative surgery or local therapy
* Patients with documented objective radiographic progression during or after local therapy or after treatment with sorafenib or lenvatinib or intolerance to or refusal to receive either agent
* Patients with at least one prior systemic therapy for HCC
* Patients eligible to be treated with nivolumab
* Patients with measurable disease based on RECIST v1.1
* Patients with Child-Pugh class A liver score within 7 days of first study dose
* Patients with no history of hepatic encephalopathy
* Patients with no prior or current clinically significant ascites as measured by physical examination and that requires active paracentesis for control (patients with ascites only on radiographic imaging are eligible)
* Patients with HBV infection must have received antiviral therapy for at least 12 weeks and HBV viral load must be documented to be <100 IU/mL within 7 days of first study dose
* Patients with no active co-infection with HBV and HCV or HBV and HDV
* Patients with no active drug or alcohol abuse

Exclusion Criteria:

* Patients with tyrosine kinase inhibitor treatment within 2 weeks of first study dose
* Patients with esophageal or gastric variceal bleeding within the past 6 months
* Patients with portal vein invasion at the main portal (Vp4) or the inferior vena cava or cardiac involvement of HCC based on imaging
* Patients with previous solid organ or hematologic transplantation
* Patients with active autoimmune disease requiring systemic treatment in the past 2 years
* Patients with diagnosis of immunodeficiency or receiving systemic steroid therapy or other immunosuppressive therapy within 7 days before first study dose
* Patients with previous locoregional therapy or major surgery to the liver within 6 weeks before first study dose
* Patients with minor surgery to liver or another site within 1 week before first study dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Through study completion, an average of 1 year
  Adverse Events evaluated according to CTC-AE

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression, assessed up to 12 months
  Partial and Complete response according to RECIST V1.1
Duration of Response (DOR) | From date of randomization until the date of first documented progression, assessed up to 12 months
Progression-Free Survival | From date of randomization until the date of first documented progression, assessed up to 24 months
Alpha Fetoprotein Serum concentrations | Every 2 weeks, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Darren SIGAL, MD, Principal Investigator — Scripps Clinic/Scripps MD Anderson Cancer Center
Locations (2):
- United States (2):
  - Scripps Clinic Torrey Pines, La Jolla, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No